CLINICAL TRIAL: NCT00133445
Title: Randomized, Single Blinded Study of the Safety and Immunogenicity of Pentavalent DTaP-Hep B-IPV Combination Vaccine (Pediarix™; GlaxoSmithKline (GSK) Biologicals) Administered to Healthy Neonates and Infants at Birth, 2, and 6 Months of Age Compared to a Routine Infant Schedule at 2, 4, and 6 Months of Age
Brief Title: Pentavalent DTaP-Hep B-IPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-062
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-10

CONDITIONS: Diphtheria; Hepatitis B; Poliomyelitis; Pertussis; Tetanus
Keywords: Pentavalent vaccine, Pediarix, DTaP-Hep B-IPV vaccine
MeSH Terms: conditions — Diphtheria; Hepatitis B; Poliomyelitis; Whooping Cough; Tetanus

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Group A (Experimental): Group A will receive DTaP-HepB-IPV (Pediarix™) vaccine along with other required vaccines at birth, 2 and 6 months of age.
  Interventions: Biological: DTaP-Hep B-IPV Vaccine; Drug: Placebo
- Group B (Active Comparator): Group B will receive the monovalent HepB vaccine (Engerix-B) at birth, the DTaP-HepB-IPV (Pediarix™) vaccine with other vaccines at 2, 4 and 6 months of age.
  Interventions: Biological: DTaP-Hep B-IPV Vaccine; Biological: Monovalent Hep B Vaccine

INTERVENTIONS:
Biological: DTaP-Hep B-IPV Vaccine — U.S. licensed 13-Dec-2002. Dosage equal to 0.5 mL administered intramuscularly. Combination vaccine.
Biological: Monovalent Hep B Vaccine — U.S. licensed monovalent hepatitis B vaccine; each 0.5 mL dose contains 10 mcg of hepatitis B surface antigen absorbed on 0.25 mg aluminum hydroxide. The vaccine is given to infants as a 0.5 mL dose intramuscularly.
  Arms: Group B
Drug: Placebo — Commercially prepared normal saline. The dose will be 0.5 mL administered intramuscularly.
  Arms: Group A

SUMMARY:
The purpose of this study is to evaluate the safety of administering a combination vaccine (DTaP-HepB-IPV; Pediarix™) to infants at birth, 2 and 6 months compared to the administration of a HepB vaccine at birth and the same combination vaccine at 2, 4, and 6 months of age. Additionally, researchers will assess the body's antibody response (proteins produced by the body's immune system that help fight infections) following each vaccine dose. The study will enroll 5 healthy newborns, ages 0-5 days. Participants will be involved in study related procedures for up to 288 days, including blood sample collection and 5 study visits.

DETAILED DESCRIPTION:
Routine immunization at birth is standard for hepatitis B in the United States (US) and for hepatitis B, polio and tuberculosis (BCG) in many countries. Other vaccines have not been routinely administered at birth largely due to concerns relating to immaturity of the neonatal immune system and the possibility of reduced immune response to vaccine antigens. With the recent licensure in the US of a pentavalent combination vaccine (DTaP-Hep B-IPV; Pediarix™) researchers propose to evaluate a new immunization schedule that includes a birth dose of this vaccine, in an effort to determine adequacy of neonatal immune response to the study vaccine antigens. The primary objectives of this study are: to evaluate the safety of administering the pentavalent combination vaccine (DTaP-HepB-IPV; Pediarix™) to infants at birth, two and six months of age compared to the administration of a hepatitis B vaccine (Engerix-B) at birth and the same pentavalent combination vaccine at two, four and six months of age; and to assess age specific antibody response following each vaccine dose. Five healthy newborns; 0 to 5 days of age, greater than or equal to 37 weeks gestation, and greater than 2500 gm birth weight were recruited from two Southern California Kaiser Permanente medical centers. Infants were randomized to one of 2 study groups: Group A received DTaP-HepB-IPV (Pediarix™) vaccine along with other required vaccines at birth, two, six months of age; Group B received the monovalent hepatitis B vaccine (Engerix-B) at birth, the DTaP-HepB-IPV (Pediarix™) vaccine with other vaccines at two, four and six months. Children will be evaluated for post-vaccination adverse events. Blood will be collected and immunogenicity evaluated by standardized humoral immunologic assays. The main outcome measures are to assess immune responses to each vaccine antigen over time, antibodies to pertussis (PT, FHA, PRN), diphtheria, tetanus, haemophilus influenzae type b (Hib), polio (Types 1, 2, 3) and hepatitis B (HbsAg). The secondary outcome measures are to assess vaccine safety, systemic and local immediate reactions.

ELIGIBILITY:
Inclusion Criteria:

Prenatal Inclusion Criteria

* Generally healthy, pregnant mother
* Mother will deliver at a Kaiser Permanente Medical Center participating in the study
* Ability of the parent(s) to understand and comply with the requirements of the protocol
* Signed informed consent by parent(s)

Birth Inclusion Criteria

* Healthy newborn 0 to 5 days of age
* Gestational age greater than or equal to 37 weeks to less than or equal to 42 weeks and birth weight greater than 2500 grams
* Signed informed consent obtained
* Mother continues to be eligible by prenatal screening criteria
* Newborn will receive future well child care at a Kaiser Permanente study clinic
* After reviewing with parent(s) the study procedures and informed consent, parent wishes to continue in the study

Exclusion Criteria:

Prenatal Exclusion Criteria

* Mother positive for hepatitis B surface antigen (HBsAg) or whose antigen status is unknown
* Mother positive for human immunodeficiency virus (HIV) or whose antigen status is unknown
* Mother positive for rapid plasma reagin (RPR) (syphilis) or whose antigen status is unknown
* Mother or immediate family member has impaired immunologic function
* Mother is expected to take immune suppressant medications during the last trimester of pregnancy
* Mother is expected to receive blood, blood products or immunoglobulin preparation (including hepatitis B immune globulin [HBIG]) during the last trimester of the pregnancy
* Mother with insulin dependent diabetes
* Mother with pre-eclampsia, eclampsia or abruptio placentae
* Pregnancy associated with known congenital defects
* Mother participating in another study with a non-Food and Drug Administration (FDA) approved drug, vaccine or device
* Parent(s)/guardian cannot be contacted by telephone
* Parent(s)/guardian will not continue well child care at a Kaiser Permanente study clinic
* Mother who is requesting that cord blood be retained for stem cell preservation
* Other maternal conditions that, in the opinion of the investigator, would interfere with the study

Birth Exclusion Criteria

* Current receipt of antibiotics for suspected infection in mother or newborn (based on presence of maternal fever greater than or equal to 38.0 degrees Celsius or prolonged rupture of membranes greater than or equal to 18 hours)
* Rectal temperature greater than or equal to 38.0 degrees Celsius
* Newborn receiving resuscitation [including intubation, mechanical ventilation or intravenous (IV) medication] at birth
* Suspected medical, congenital, developmental or surgical disease, including immunodeficiency, neurology disorder or seizure disorder, severe congenital anomalies or multi-organ dysfunction
* Prior receipt of hepatitis B vaccine or any other vaccine
* Received or plans to receive any immunosuppressant medication
* Receipt of blood products or immunoglobulin [including Hepatitis B Immune Globulin (HBIG)]
* Clinically significant findings on review of medical history and physical exam determined by the investigator or sub-investigator to be sufficient for exclusion
* Mother of newborn with insulin dependent diabetes
* Mother of newborn with pre-eclampsia, eclampsia or abruptio placentae
* Mother of newborn positive for HBsAG, HIV or RPR (syphilis) or whose antigen status is unknown
* Impaired immunologic function in newborn or family member
* Any condition determined by the investigator that would interfere with the evaluation of the vaccine or be a potential health risk to the subject
* Newborn is participating in another research study or has received a non-FDA approved drug or vaccine (excluding formula preparations) prior to study entry
* Parent(s)/guardian who are unable to be contacted by telephone

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2005-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To assess the immune responses to each vaccine antigen over time, antibodies to pertussis (PT, FHA, PRN), diphtheria, tetanus, Hib, polio (Types 1, 2, 3) and hepatitis B (HbsAg) will be evaluated. | Day 0-5, Day 53-70, Day 113-130, Day 173-190, and Visit 4 + (28-42 days).

SECONDARY OUTCOMES:
To assess vaccine safety, systemic and local immediate reactions. | 30 mins after each immunization; 7 days following each vaccination; contacted 2-3 and 8 days following each vaccination to collect AE information; SAEs will be collected throughout study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center For Vaccine Research, Torrance, California, United States